CLINICAL TRIAL: NCT07024732
Title: An Open-label Single Ascending Dose Safety and Tolerability Clinical Trial of PST-611 in Subjects With Dry Age-related Macular Degeneration
Brief Title: A Safety and Tolerability Clinical Trial of PST-611 in Dry Age-related Macular Degeneration
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eyevensys (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PST-611-CT1; 2024-519025-37-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-05; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Dry Age Related Macular Degeneration
Keywords: Dry Age Related Macular Degeneration; PST-611

STUDY DESIGN:
Intervention Model Description: Single ascending dose design with 2 sequential dose groups (low dose group followed by high dose group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active treatment (Experimental): This arm consists of 2 dose groups receiving a single ascending dose of PST-611. These groups will be dosed sequentially, low dose followed by high dose.
  Interventions: Biological: PST-611

INTERVENTIONS:
Biological: PST-611 — PST-611 is a naked plasmid DNA encoding human transferrin administered into the ciliary muscle

SUMMARY:
The goal of this interventional study is to evaluate the safety and tolerability of single ascending doses of PST-611 in men and women over the age of 50 with dry age-related macular degeneration (AMD).

The main question it aims to answer is: Is PST-611-CT1 safe for participants?

Participants will:

* Receive a single dose of PST-611
* Will be followed up for a total of 16 weeks following PST-611 administration

DETAILED DESCRIPTION:
The maximum study duration per patient is 28 Weeks (including an up to 12 week screening period + 16 weeks of follow-up after treatment).

The study is a single ascending dose study that investigates two PST-611 dose levels (low and high doses) in 2 successive dose groups. The study will enroll up to 12 participants.

ELIGIBILITY:
Inclusion Criteria:

Subjects must give written informed consent, be able to make the required trial visits and follow instructions.

Female and male subjects must be 50 years of age or older. Female subjects of childbearing potential must not be pregnant or breast-feeding and must have a negative urine pregnancy test at baseline and throughout the study. They must agree to practice at least one effective method of birth control following administration of study medication.

In the study eye, at least one of the following must be present at OCT and attributed to AMD, as evaluated by the Investigator: Incomplete RPE and Outer Retinal Atrophy (iRORA), or Complete RPE and Outer Retinal Atrophy (cRORA).

Best-Corrected Visual Acuity (BCVA), must be 23 ETDRS letters (approximate Snellen equivalent 20/320) or better in the study eye.

Subject's fellow eye BCVA must be 34 letters (approximate Snellen equivalent 20/200) or better.

Exclusion Criteria:

Both eyes: any active intraocular or periocular infection or inflammation (eg, infectious blepharitis, infectious conjunctivitis, keratitis, scleritis, endophthalmitis), or history of intraocular or periocular infection or inflammation in the 12 weeks (84 days) prior to the PST-611 administration.

Study eye: Any intraocular surgery (including cataract surgery) or intravitreal (IVT) or periocular corticosteroid injection within 12 weeks (84 days) prior to the PST-611 administration.

Study eye: Any anti-VEGF IVT treatment within 4 weeks (28 days) prior to PST-611 dosing OR subjects who have required and received regular monthly injections of anti-VEGF drugs in the months preceding the trial and would thus have a higher likelihood of requiring and anti-VEGF treatment within 28 days of the PST-611 administration.

Study eye: media opacity that interferes with fundus imaging or is likely to require surgery during the trial period.

Study eye: subject with history of glaucoma filtering surgery (e.g. trabeculectomy or aqueous shunt implant) or who underwent eye surgery within 12 weeks (84 days) of the PST-611 administration. Study eye: subject who has uncontrolled intraocular pressure of ≥ 25 mmHg in the SE at the screening and baseline visits.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Screening to week 16
  Ocular and non-ocular adverse events frequency and severity

SECONDARY OUTCOMES:
Intraocular pressure | Screening to Week 16
  Intraocular pressure measured in mmHg
Best corrected visual acuity | Screening to Week 16
  Best corrected visual acuity measured in ETDRS letters
Slit lamp biomicroscopy examination | Screening to Week 16
  Abnormal examination results will be recorded
Dilated ophthalmoscopy examination | Screening to Week 16
  Abnormal examination results will be recorded
Color fundus photography | Screening to Week 16
  Abnormal findings will be recorded
Spectral Domain-Optical Coherence Tomography | Screening to Week 16
  Abnormal findings will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Karine Bigot, PhD, Study Director — PulseSight Therapeutics
Locations (2):
- France (2):
  - CHU de Grenoble-Hôpital Michallon, Grenoble
  - Hôpital Cochin, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bigot K, Gondouin P, Benard R, Montagne P, Youale J, Piazza M, Picard E, Bordet T, Behar-Cohen F. Transferrin Non-Viral Gene Therapy for Treatment of Retinal Degeneration. Pharmaceutics. 2020 Sep 1;12(9):836. doi: 10.3390/pharmaceutics12090836. PMID 32882879